CLINICAL TRIAL: NCT01336907
Title: Comparison Between Home Macular Perimeter and OCT Visual Field Defects in Patients With CNV
Brief Title: Comparison Between Home Macular Perimeter and Optical Coherence Tomography (OCT) Visual Field Defects in Patients With Choroidal Neovascularization (CNV)
Status: Withdrawn | Type: Observational
Why Stopped: never started
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Sponsor
Organization: Notal Vision Inc. (Industry)
Other Study IDs: HMP-DTR-01
Record Dates: First submitted 2011-04-13; First posted 2011-04-18 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Age Related Macular Degeneration; Choroidal Neovascularization
Keywords: CNV; AMD; Wet-treated CNV
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- naive CNV subjects: Newly diagnosed CNV, before any treatment (naïve)
- previously diagnosed CNV subjects: Previously diagnosed CNV if last treatment is older than 4 months (reactivated)

SUMMARY:
The FORESEE HOME is intended for the early detection of central and paracentral irregularities (abnormalities) in the visual field, most commonly associated with Age Related Macular Degeneration (AMD). However, the device has the ability to detect the development of the lesion post treatment and therefore to assess in determination of the next treatment.

The Optical Coherence Tomography (OCT) may be used as well to identify choroidal neovascularization (CNV). Comparison between the two methods will allow better understanding of both devices.

The FORESEE HOME can be used as an assessment tool for the progression and success of the treatment given to AMD lesions. Therefore, evaluating the size and the location of the treated lesions may serve as an additional tool.

ELIGIBILITY:
Inclusion Criteria:

* For naïve CNV lesion - diagnosed in less than 60 days. OR For re-activated CNV lesion - treated more than 4 month from the diagnosis.

  * Intent to treat the study eye (SE)
  * Corrected VA better than 6/45 (20/150) in SE
  * Subject is capable and willing to sign a consent form and participate in the study
  * Age > 55 years
  * Subject declared that he or she knows how to operate a computer mouse

Exclusion Criteria:

* Evidence of macular disease other than AMD or glaucoma in SE
* Presence of any significant media opacity that precludes a clear view of the macular area as identified in the SE by biomicroscopy
* Any ocular surgery performed within 3 months prior to study entry in the SE * Participation in another study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CNV subjects
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Investigate the correlation between features of CNV lesions as measured with SD OCT and in the ForeseeHome. | 3-4 months
  the measures are Height of Pigment Epithelial Detachment , Sub Retinal Fluid Thickness , Maximum Diameter of Largest Retinal Cyst , Maximum Retinal Thickness , Central Retinal Thickness

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Querques, Dr., Principal Investigator — Department of Ophthalmology, Centre Hospitalier Intercommunal de Creteil, University Paris XII, Paris, France
Locations (1):
- Centre Hospitalier Intercommunal de Creteil, Paris, France

REFERENCES:
- See also: sponsor's site — http://www.notalvision.com